CLINICAL TRIAL: NCT04559646
Title: Application of the Haemostatic Solution "Haemoblock" to Reduce the Risk of Pacemaker Pocket Hematoma
Brief Title: Application of the "Haemoblock" in Pacemaker Patients
Status: Completed | Type: Observational
Sponsor: Ryazan State Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: PEGASUS2020
Record Dates: First submitted 2020-09-16; First posted 2020-09-23 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Hematoma Postoperative
Keywords: Cardiac implantable electronic devices; Pacing; Pocket hematoma; Haemorrhagic complications
MeSH Terms: interventions — Blood Specimen Collection; Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A "Haemoblock": 100 patients. Haemostatic solution "Haemoblock" will be used after pocket formation during pacemaker implantation.
  Interventions: Procedure: Pacemaker implantation; Drug: Haemostatic solution "Haemoblock" application; Diagnostic Test: Ultrasound of pacemaker pocket; Diagnostic Test: Blood sampling; Diagnostic Test: Echocardiography
- Group B "Control": 100 patients. Saline solution will be used after pocket formation during pacemaker implantation.
  Interventions: Procedure: Pacemaker implantation; Drug: Saline solution application; Diagnostic Test: Ultrasound of pacemaker pocket; Diagnostic Test: Blood sampling; Diagnostic Test: Echocardiography

INTERVENTIONS:
Procedure: Pacemaker implantation — Implantation of the pacemaker due to indications in patients with atrioventricular block, sick sinus syndrome, atrial fibrillation with impaired atrioventricular conduction or other.
Drug: Haemostatic solution "Haemoblock" application — Haemostatic solution "Haemoblock" will be used after pocket formation during pacemaker implantation.
  Other Names: "Haemoblock" application
  Groups: Group A "Haemoblock"
Drug: Saline solution application — Saline solution will be used after pocket formation during pacemaker implantation.
  Other Names: Saline application
  Groups: Group B "Control"
Diagnostic Test: Ultrasound of pacemaker pocket — Pacemaker pocket ultrasound examination to diagnose pocket hematoma 3-5 days after surgery.
Diagnostic Test: Blood sampling — Blood sampling for Platelet, Prothrombin, Fibrinogen, International Normalized Ratio, Creatinine, Albumin evaluation.
Diagnostic Test: Echocardiography — Heart ultrasound examination for left ventricular ejection fraction measurement.

SUMMARY:
Pocket hematoma is a known complication of pacemaker (PM) implantation. Pocket hematoma is accompanied by a local discomfort associated with the infiltration of subcutaneous tissue. In some cases, this complication requires repeated surgical revisions, which increases the risk of infection, and increases the duration of a hospital stay. The search for ways to prevent bleeding from the PM pocket is of great practical interest. This question is especially acute in relation to patients who are constantly on anticoagulation and/or antiplatelet therapy. A number of authors propose to carry out complete or partial cancellation of these drugs for the period before surgery and in the early postoperative period. In our opinion, this approach in most cases carries a potential risk to the health of patients, especially in the case of patients who have previously undergone surgical correction of valve insufficiency and/or who have undergone percutaneous endovascular interventions.

The use of local hemostatic drugs is one of the promising directions for increasing the efficiency of intraoperative hemostasis. The haemostatic solution "Haemoblock" has shown its hemostatic potential in general surgical practice. The possibilities of "Haemoblock" in the prevention of pocket hematoma have not been studied. The hemostatic effect of "Haemoblock" is achieved within 1-2 minutes due to the formation of a clot with blood plasma proteins, first of all with albumin. As a result of the action of the "Haemoblock", a strong polymethacrylate membrane is formed on the surface of the wound, which, among other things, has a bactericidal effect.

DETAILED DESCRIPTION:
А multicenter research trial will be conducted at 6 medical centers:

* Ryazan State Medical University (Ryazan);
* Federal State Budgetary Institution "Federal Center for Cardiovascular Surgery" of the Ministry of Health of the Russian Federation (Astrakhan);
* Federal State Budgetary Institution "Federal Center for Cardiovascular Surgery" of the Ministry of Health of the Russian Federation (Penza);
* Federal State Budgetary Institution "Federal Center for Cardiovascular Surgery" of the Ministry of Health of the Russian Federation (Chelyabinsk);
* Federal State Budgetary Institution "Federal Center for Cardiovascular Surgery" of the Ministry of Health of the Russian Federation (Kaliningrad);
* Federal State Budgetary Institution "Federal Center for Cardiovascular Surgery" of the Ministry of Health of the Russian Federation (Khabarovsk).

Haemostatic solution "Haemoblock" provided by Autonomous non-profit organization "MOSCOW REGIONAL SCIENTIFIC RESEARCH INSTITUTE OF BLOOD".

The study will include 200 patients with indications for pacemaker implantation (atrioventricular block, sick sinus syndrome, atrial fibrillation with impaired atrioventricular conduction or other).

Before starting the study, the patient must give written consent to participate in this study after familiarizing him with the purpose and rules of the clinical study.

All patients during randomisation will be divided into 2 groups:

Group A "Haemoblock" - 100 patients. Haemostatic solution "Haemoblock" will be used after pocket formation during pacemaker implantation (sterile gauze swabs are soaked in 15 ml of "Haemoblock" solution and applied in pacemaker pocket, then pacemaker pocket will be irrigated with 5 ml of "Haemoblock" solution without rinsing).

Group B "Control" - 100 patients. Same procedure will be performed with saline solution in this group.

Before surgery blood sampling, echocardiography will be performed in all patients.

3-5 days after surgery ultrasound of pacemaker pocket will be performed in all patients.

The observation period for patients will be 30 days.

ELIGIBILITY:
Inclusion Criteria:

* availability of informed consent of the patient to participate in the study;
* men and women aged 40-85 years with indications for pacemaker implantation, taking oral anticoagulants before surgery for at least 7 days;

Exclusion Criteria:

* hypoalbuminemia;
* known contraindications for the study haemostatic solution "Haemoblock";
* severe arterial hypertension: Systolic blood pressure ≥ 200 mmHg and/or Diastolic blood pressure ≥ 110 mmHg;
* unstable forms of ischemic heart disease;
* hemostasis disorders in the number of platelets, prothrombin, fibrinogen levels, or International Normalised Ratio above 3.0
* LVEF according to Simpson <35%;
* the period of pregnancy and lactation;
* chronic renal failure: creatinine clearance less than 40 ml/min;
* hemoglobin level <90 g/l;
* participation in another study.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 patients with indications for pacemaker implantation (atrioventricular block, sick sinus syndrome, atrial fibrillation with impaired atrioventricular conduction or other).
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
The presence of free fluid (blood) in the pacemaker pocket in the early postoperative period, diagnosed by ultrasound. | Up to 30 days after pacemaker implantation.
  Ultrasound of pacemaker pocket to diagnose pocket hematoma will be performed in all patients. The presence of a hematoma (fluid) in the pacemaker pocket before the ultrasound can be verified after examination by the surgeon by the detection of palpable infiltration, smoothing the pacemaker contour, the presence of a fluctuation effect.

SECONDARY OUTCOMES:
Drainage installation during surgery. | During surgery.
  Installation of a drainage system during pacemaker implantation for draining hematoma after surgery.
Hematoma drainage duration. | Up to 7 days after pacemaker implantation.
  Duration of hematoma drainage after pacemaker implantation if installed during surgery.
Imbibition of soft tissues near pacemaker pocket. | Up to 30 days after pacemaker implantation.
  Imbibition of soft tissues around pacemaker pocket detected on physical examination.
Exceeding the average length of hospital stay. | Up to 30 days after pacemaker implantation.
  Exceeding the average length (7 days) of hospital stay.
Pacemaker implantation complications and cardiac events (stroke, transient ischemic attack, bleeding, pericarditis, cardiac tamponade, infection). | Up to 30 days after pacemaker implantation.
  Pacemaker implantation complications and cardiac events (stroke, transient ischemic attack, bleeding, pericarditis, cardiac tamponade, infection) development during observation period.

CONTACTS AND LOCATIONS:
Overall Officials: Igor A. Suchkov, MD, DSc, Principal Investigator — Ryazan State Medical University
Locations (1):
- Ryazan State Medical University, Ryazan, Ryazan Oblast, Russia

IPD SHARING:
Plan to Share IPD: Undecided
Basic demographic data, including sex, age, and ethnicity are to be shared if allowed by the privacy policy.